CLINICAL TRIAL: NCT00486369
Title: SMC021A - Absorption, Efficacy and Tolerance in Patients With Osteoarthritis. A Placebo-Controlled 14-Days Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nordic Bioscience A/S (Industry)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSMC021C2102
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2007-06

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, oral salmon calcitonin, tolerability, biomarkers
MeSH Terms: conditions — Osteoarthritis | interventions — salmon calcitonin

INTERVENTIONS:
Drug: Oral salmon calcitonin

SUMMARY:
The purpose of this study is to expose patients with OA to calcitonin and to determine plasma calcitonin levels after administration of 0.6 mg and 0.8 mg oral calcitonin. Also the purpose is to assess the effect of different doses of oral calcitonin (0.6 mg and 0.8 mg oral) compared to placebo on serum CTX-I and CTX-II. Finally to assess the tolerance profile of different doses/formulations of oral calcitonin compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Medical history and symptoms of knee osteoarthritis

Exclusion Criteria:

* Any other disease or medication affecting the bone or cartilage.
* Any clinical signs or laboratory evidence diseases, which in the Investigator's opinion would preclude the participant from adhering to the Protocol or completing the trial.

Ages: 52 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-01

SECONDARY OUTCOMES:
Changes in Urine CTX-I and CTX-II
Changes in serum osteocalcin and serum CTX-I
Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bente J Riis, M.D., Study Chair — Nordic Bioscience A/S
Locations (1):
- CCBR A/S, Ballerup Municipality, Denmark

REFERENCES:
- [Derived] Karsdal MA, Byrjalsen I, Bay-Jensen AC, Henriksen K, Riis BJ, Christiansen C. Biochemical markers identify influences on bone and cartilage degradation in osteoarthritis--the effect of sex, Kellgren-Lawrence (KL) score, body mass index (BMI), oral salmon calcitonin (sCT) treatment and diurnal variation. BMC Musculoskelet Disord. 2010 Jun 17;11:125. doi: 10.1186/1471-2474-11-125. PMID 20565725
- [Derived] Karsdal MA, Byrjalsen I, Henriksen K, Riis BJ, Lau EM, Arnold M, Christiansen C. The effect of oral salmon calcitonin delivered with 5-CNAC on bone and cartilage degradation in osteoarthritic patients: a 14-day randomized study. Osteoarthritis Cartilage. 2010 Feb;18(2):150-9. doi: 10.1016/j.joca.2009.08.004. Epub 2009 Sep 1. PMID 19747581